CLINICAL TRIAL: NCT05081739
Title: Donor-Derived Cell-free DNA to DETect REjection in Cardiac Transplantation
Acronym: DETECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor made decision to pause study while it was still in development phase. The FDA and IRB approval process had not been completed. No sites were activated. No subjects had been recruited for this study.
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-053-TRP
Record Dates: First submitted 2021-09-17; First posted 2021-10-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Heart Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospera Surveillance (Experimental): Subjects will undergo Prospera testing in accordance with the institution's Control Group EMB surveillance standard of care schedule, which is expected to be approximately every other week months 2 and 3, then monthly through months 4 through 6, then every 1-3 months during months 7 through 12. Prospera test results will be provided to investigators. Prospera cfDNA level < 0.15 % will be interpreted as negative, and screening EMB will be omitted. EMB will be performed for cfDNA level ≥ 0.15 %. At any time, the clinical team may perform for cause EMB for standard clinical indications (e.g., evidence of graft failure) as per the treating team's discretion.
  Interventions: Diagnostic Test: Prospera Transplant Assessment
- EMB Surveillance (Active Comparator): Subjects will undergo surveillance EMB per the institution's standard clinical care, which is expected to be approximately every other week months 2 and 3, then monthly through months 4 through 6, then every 1-3 months during months 7 through 12. At any time, the clinical team may perform for cause EMB for standard clinical indications (e.g., evidence of graft failure) as per the treating team's discretion.
  Interventions: Procedure: Endomyocardial biopsy

INTERVENTIONS:
Diagnostic Test: Prospera Transplant Assessment — Prospera™ detects allograft rejection noninvasively and with high accuracy by measuring the fraction of dd-cfDNA in the patient's blood, without the need for prior donor or recipient genotyping.
  Prospera is a commercially available LDT developed by Natera, Inc. Natera is a laboratory certified under the Clinical Laboratory Improvement Amendments (CLIA).
  Arms: Prospera Surveillance
Procedure: Endomyocardial biopsy — Subjects will undergo surveillance EMB per the institution's standard clinical care, which is expected to be approximately every other week in months 2 and 3, then monthly through month 6, then every 1-3 months through the end of month 12.
  Arms: EMB Surveillance

SUMMARY:
The study objective is to demonstrate that rejection surveillance of heart transplant recipients with Prospera dd-cfDNA is non-inferior to rejection surveillance with endomyocardial biopsy and histology in the first post-transplant year.

DETAILED DESCRIPTION:
Subjects will be enrolled into the study while on the transplant waiting list prior to heart transplantation. All subjects will follow the center's standard of care surveillance schedule from transplant through 4 weeks post-transplantation. EMB during this phase is expected to occur roughly weekly.

Subjects will be randomized in a 1:1 ratio 30 days (± 7 days) post-transplant to Prospera surveillance (Study Group) versus EMB surveillance (Control Group, standard clinical care). Rejection surveillance (Prospera testing in the Study Group and EMB in the Control Group) will be performed at times corresponding to the institutional standard of care schedule for rejection surveillance.

Study Group: Prospera Surveillance (300 Subjects) Subjects will undergo Prospera testing at times corresponding to the institution's graft surveillance schedule. Prospera test results will be provided to the clinical team. Prospera cfDNA level < 0.15% will be interpreted as negative and a surveillance EMB will be omitted. Prospera cfDNA ≥ 0.15% will be followed by EMB. A for-cause EMB can be done per the clinical team's discretion at any time.

Control Group: EMB Surveillance (standard of care) (300 Subjects) Subjects will undergo surveillance EMB per the institution's standard clinical care.

The study intervention will be during the first 12 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older at the time of signing informed consent.
2. On the heart transplant waiting list and expected to receive a heart transplant.
3. Able to read, understand and provide written informed consent.
4. Able and willing to comply with the study visit schedule, study procedures and study requirements.

Exclusion Criteria:

1. Heart transplantation has been performed.
2. Concurrent multiple solid organ or tissue transplant
3. Prior history of any organ or cellular transplantation.
4. Planned use of other commercially available or investigational cfDNA or gene expression profile assays.
5. Pregnant.
6. Hemodynamically unstable or other serious medical condition that may adversely affect the subject's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the use of Prospera for post-transplant surveillance is non-inferior to the current standard of care, EMB surveillance, with respect to the primary composite endpoint. | 12 months
  The primary endpoint of the study is a composite endpoint defined as the first occurrence of one or more of the following events after transplant:
  1. Treated rejection with or without graft dysfunction and/or graft dysfunction requiring treatment with pulse dose steroids, monoclonal antibodies, plasmapheresis, and/or intravenous immunoglobulin (IVIg)
  2. Graft dysfunction
  3. Re-transplantation
  4. Death
  Clinical endpoints are defined as follows:
  * Rejection: ISHLT ACR Grade ≥ 2R or AMR Grade ≥ pAMR1
  * Graft dysfunction: LVEF decline >10% from baseline and < 50% absolute LVEF by echocardiography
  * Re-transplantation: being listed for re-transplant or being re-transplanted

CONTACTS AND LOCATIONS:
Overall Officials: Michael Olymbios, MD, Study Director — Natera, Inc.; Palak Shah, MD, Principal Investigator — Inova Health Care Services; Josef Stehlik, MD, Study Chair — University of Utah